CLINICAL TRIAL: NCT06972056
Title: A Comparative Effectiveness Study of Oral Medications Used for Migraine Prevention: The APT Comparison Study
Brief Title: Comparative Effectiveness of Migraine Preventive Medications: The APT Comparison Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Iowa (Other); Patient-Centered Outcomes Research Institute (Other); AbbVie (Industry)
Responsible Party: Principal Investigator, Todd J. Schwedt, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-012753; MI-2023C2-33021 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-08

CONDITIONS: Migraine
Keywords: Migraine; Migraine with aura; Migraine prevention
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura | interventions — atogepant; Propranolol; Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Atogepant (Active Comparator): Participants who are randomized to this arm will take up to 60mg daily for 12 weeks.
  Interventions: Drug: Atogepant 60 mg
- Propranolol (Active Comparator): Participants randomized to this arm will take up to 160 mg daily for 12 weeks.
  Interventions: Drug: Propranolol 160 mg
- Topiramate (Active Comparator): Participants randomized to this arm will take up to 100 mg daily for 12 weeks .
  Interventions: Drug: Topiramate 100 mg

INTERVENTIONS:
Drug: Atogepant 60 mg — Atogepant at a dose up to 60 mg daily.
  Other Names: Qulipta
  Arms: Atogepant
Drug: Propranolol 160 mg — Daily propranolol up to 80 mg twice daily.
  Other Names: Inderal
  Arms: Propranolol
Drug: Topiramate 100 mg — Daily topiramate, up to 50 mg twice daily
  Other Names: Topamax
  Arms: Topiramate

SUMMARY:
This goal of this study is to compare three medications used for migraine preventive treatment.

This study will compare atogepant, a newer migraine preventive medication, with two older preventive medications, topiramate and propranolol. It will be determined if one works better and is more tolerable than the others.

Research participants will:

* Be randomly assigned to one of the three medications.
* Provide information about their migraine pattern using a daily headache diary and during research visits.

DETAILED DESCRIPTION:
This is a prospective, randomized, comparative effectiveness clinical trial of atogepant, propranolol, and topiramate for the prevention of migraine in adults.

Eligible participants will provide information in a daily headache diary for four weeks. If after those four weeks they are still eligible for the study, they will be randomized to one of the study medications and receive study medication for twelve weeks.

Research visits occur at baseline, four weeks later for the randomization visit, and then at post-randomization weeks four, eight, twelve, twenty-four, and forty-eight.

Participants provide data using a headache diary (first 16 weeks of the study) and during research visits.

The primary endpoint is the proportion of participants in each treatment group who are "treatment responders" defined as completing the first twelve weeks of the study on the assigned medication and having a 50% or greater reduction in moderate severe headache days during weeks 9-12 post-randomization compared to the four weeks pre-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-70 years of age at the time of enrollment
* Migraine with aura, migraine without aura, and/or chronic migraine; according to ICHD-3 diagnostic criteria. (Those with daily or continuous headaches are not excluded.)
* Migraine onset prior to 50 years of age
* Migraine present for at least 12 months at the time of enrollment
* At least four "moderate to severe headache days" per month (by patient self-report and then confirmed during four-week pre-randomization headache diary phase) A "moderate to severe headache day" is defined as a day during which there is a headache of moderate to severe intensity that lasts for at least four hours, or a day on which a migraine-specific acute medication is taken to treat headache.
* If already taking a migraine preventive treatment, willing to continue with that treatment without dose change during the first 16 weeks of the study, including the 4-week run-in phase and 12-week randomized phase.
* Not pregnant or breastfeeding
* Women of childbearing potential must agree to use effective methods of contraception to reduce the risk of pregnancy.
* Willingness and ability to provide informed consent.
* Willingness and ability to complete all research visits.

Exclusion Criteria:

* Contraindications to taking atogepant, propranolol, or topiramate.
* Currently taking atogepant, propranolol, or topiramate*
* Previously took atogepant, propranolol, or topiramate*
* Unwillingness to take atogepant, topiramate, or propranolol.
* Current use of a CGRP-targeting preventive medication or beta-blocker
* Migraine with brainstem aura
* Hemiplegic migraine
* Retinal migraine
* Migraine aura without headache (exclusively)
* Pure menstrual migraine
* Trigeminal autonomic cephalalgias
* Facial neuralgias
* Secondary headache disorders (medication overuse headache is not an exclusion)
* Migraine preventive treatment has been started or dose has been changed within 12 weeks prior to potential enrollment.
* Used opioids or butalbital on five or more days per month on average for at least 3 months prior to enrollment.
* Current or past epilepsy
* Severe hepatic impairment
* Moderate or more severe renal impairment * Occasional as needed use of propranolol, currently or in the past, is not an exclusion, such as taking as needed propranolol for treatment of anxiety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1335 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Responder (atogepant vs. topiramate; atogepant vs. propranolol) | Weeks 9-12 post-randomization compared to the 4 weeks prior to randomization
  This study will use a "treatment responder" primary endpoint that will investigate medication superiority using a combination of headache frequency reduction and medication persistence. To achieve this, a binary endpoint of treatment response will be used that combines effectiveness and medication persistence at the individual level, with success defined as:
  1. Completing the first 12 weeks of the study on the assigned medication without discontinuation due to any reason, AND
  2. Having a 50% or greater reduction in moderate to severe headache days during weeks 9-12 compared to a 4-week pre-randomization period.

SECONDARY OUTCOMES:
Migraine Specific Quality-of-Life - Role Function-Restrictive | Week 12 post-randomization vs. baseline
  The role function-restrictive domain of the Migraine Specific Quality of Life questionnaire is a 7-item valid measure of functional impact of migraine on work or daily activities, relationships with family and friends, leisure time, productivity, concentration, energy, and tiredness during the past four weeks.
Treatment Responder (propranolol vs. topiramate) | Weeks 9-12 post-randomization vs. the 4 weeks prior to randomization
  This study will use a "treatment responder" primary endpoint that will investigate medication superiority using a combination of headache frequency reduction and medication persistence. To achieve this, a binary endpoint of treatment response will be used that combines effectiveness and medication persistence at the individual level, with success defined as:
  1. Completing the first 12 weeks of the study on the assigned medication without discontinuation due to any reason, AND
  2. Having a 50% or greater reduction in moderate to severe headache days during weeks 9-12 compared to a 4-week pre-randomization period.
Headache Impact Test-6 (HIT-6) | week 12 post-randomization vs. baseline
  The HIT-6 is a six-item questionnaire that measures the impact headaches have on a person's ability to function on the job, at home, at school, and in social situations.
Medication-Related Adverse Events | All 12 weeks of the randomized treatment phase
  This medication-related adverse event outcome will consist of all adverse events that are deemed to be at least possibly related to the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Todd J Schwedt, M.D., Principal Investigator — Mayo Clinic
Locations (17):
- United States (17):
  - Northern Arizona Healthcare, Flagstaff, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - USC Keck, Los Angeles, California
  - Clinical Research Institute, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Apple Med Research, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Washington University St Louis, St Louis, Missouri
  - Advanced Research Institute Reno, Reno, Nevada
  - JFK Neuroscience Institute, Edison, New Jersey
  - Wake Forest University Health, Winston-Salem, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Advanced Research Institute, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Advanced Research Institute Ogden, Ogden, Utah
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
As per PCORI data sharing policy
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Summer 2030 (anticipated)
Access Criteria: Per PCORI data sharing policy